CLINICAL TRIAL: NCT00706537
Title: A Multiple Dose, Randomized, Double-Blind (3rd Party Open), Placebo-Controlled Phase 1 Study To Evaluate The Pharmacokinetics And Safety Of CP-945598 In Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Phase 1 Pharmacokinetic Study Of CP-945598 In Patients With NASH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: A5351053
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2008-11

CONDITIONS: Non-Alcoholic Steatohepatitis(NASH)
Keywords: Pharmacokinetic safety NASH patients
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CP-945598 20 mg (Experimental)
  Interventions: Drug: Active treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active treatment — 20 mg CP-945598 as 15 and 5 mg tablet once daily for 3 weeks
  Arms: CP-945598 20 mg
Drug: Placebo — Placebo as two tablets once daily for three weeks
  Arms: Placebo

SUMMARY:
CP-945598 is a potent and selective Cannabinoid-1 (CB1) receptor antagonist currently being developed for the treatment of obesity. CP-945598 is also being considered as a potential treatment for non-alcoholic steatohepatitis (NASH). This study will investigate the steady-state safety, toleration and pharmacokinetics of multiple oral dose administration of CP-945598. Results will be used to estimate the pharmacokinetic characteristics in NASH patients and underwrite the safety of this compound prior to any further studies in NASH patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 25 to 40 kg/m2
* Subjects with biopsy evidence of NASH in the 2 years prior to the screening visit.

Hemoglobin ≥11 g/dL, platelet count ≥100,000 cells/mm3, neutrophil count ≥1,500cells/mm3.

Exclusion Criteria:

* Other forms than NASH liver disease.
* Decompensated or severe liver disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Urine 6-β-hydroxycortisol:cortisol ratio | 3 weeks
Adverse event monitoring, physical examinations, sitting vital sign measurements (blood pressure and pulse rate), 12-lead ECGs, laboratory safety assessments. | 8 weeks
PK for CP-945598 and its primary circulating metabolite | 6 weeks

SECONDARY OUTCOMES:
Breath ID® tests (methacetin and octanoate) | 6 weeks
Soluble and exploratory biomarkers | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Durham, North Carolina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351053&StudyName=Phase%201%20Pharmacokinetic%20Study%20Of%20CP-945598%20In%20Patients%20With%20NASH